CLINICAL TRIAL: NCT06902116
Title: Comparison of Outcome of Three Days Bowel Preparation vs No Bowel Preparation in Patients of Colostomy Reversal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Aziz Ahmad Chattha, Senior Registrar, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1038/CH-UCHS
Record Dates: First submitted 2025-02-13; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Colostomy - Stoma; Bowel Preparation; BOWEL ANASTOMOSIS

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Colostomy Reversal (Active Comparator): Patients in this group will not receive any mechanical bowel preparation prior to undergoing colostomy reversal.
  Interventions: Procedure: No Mechanical Bowel Preparation
- Group B Colostomy Reversal (Active Comparator): Patients in this group will receive 3 days bowel preparation prior to undergoing colostomy reversal.
  Interventions: Procedure: Mechanical Bowel Preparation

INTERVENTIONS:
Procedure: No Mechanical Bowel Preparation — In this group patients will not receive any mechanical bowel preparation prior to undergoing colostomy reversal.
  Arms: Group A Colostomy Reversal
Procedure: Mechanical Bowel Preparation — In this group patients will receive 3 days mechanical bowel preparation prior to undergoing colostomy reversal.
  Arms: Group B Colostomy Reversal

SUMMARY:
The goal of this trial is to compare the outcomes of colostomy reversal with three days bowel preparation with no bowel preparation in terms of anastomotic leakage, surgical site infection and hospital stay.

The important question this trial aims to answer is:

1. is there any difference in outcomes after colostomy reversal with three days gut preparation pre-operatively vs no gut preparation?

This prospective Randomized Controlled trial will include children with colostomy divided into two groups:

Group A: No Mechanical Bowel Preparation Group B: 3 Days Mechanical Bowel Preparation Participants of Group A will be admitted 1 day prior to surgery date as they require no special preparation before surgery. They will be made Nil per oral 6 hours prior to surgery. Group B participants will be admitted 3 days prior to surgery. These participants will be restricted to fiber rich diet and milk 72 hours prior to surgery. They will be shifted to clear liquids 24 hours prior to surgery. Normal saline enema will be given 8 hourly through the stoma as well as per rectally by the trained person.

Comparative outcomes will be:

1. Anastomotic leakage
2. Hospital Stay
3. Wound infection

ELIGIBILITY:
Inclusion Criteria:

* Children with colostomy between 1-15 years of age

Exclusion Criteria:

* Malnourished
* Previous history of colostomy site anastomotic leakage

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leakage | 5-10 days post operatively.
  In this outcome measure, it will be seen if there is any difference in both intervention in terms of number of participants with anastomotic (part of gut where two separate ends of colon have been sutured with each other) leakage.
Wound infection | At 7 days after surgery and then at 30 days after surgery.
  In this outcome variable, number of participants with infection at the site of colostomy reversal wound will be compared between both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Child Health Sciences, The Children's Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication after deidentification (text, table, figures and appendices)
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal in order to achieve the aims mentioned in the approved proposal. Proposals should be directed to email : azizchattha@hotmail.com

REFERENCES:
- [Background] Cavusoglu YH, Karaman A, Afsarlar CE, Karaman I, Erdogan D, Ozguner IF. Ostomy Closures in Children: Variations in Perioperative Care Do Not Change the Outcome. Indian J Surg. 2015 Dec;77(Suppl 3):1131-6. doi: 10.1007/s12262-015-1212-0. Epub 2015 Jan 19. PMID 27011524
- [Background] Ares GJ, Helenowski I, Hunter CJ, Madonna M, Reynolds M, Lautz T. Effect of preadmission bowel preparation on outcomes of elective colorectal procedures in young children. J Pediatr Surg. 2018 Apr;53(4):704-707. doi: 10.1016/j.jpedsurg.2017.03.060. Epub 2017 Mar 30. PMID 28433362

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT06902116/Prot_SAP_000.pdf